CLINICAL TRIAL: NCT02614612
Title: A Randomized, Parallel-Cohort Phase 1 Study of Itacitinib in Combination With Corticosteroids for the Treatment of Acute Graft Versus Host Disease
Brief Title: Study of Itacitinib in Combination With Corticosteroids for the Treatment of Acute GVHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-108
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Acute Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — itacitinib; INCB039110; Prednisone; Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itacitinib (200 mg) (Experimental): Itacitinib (200 mg) + prednisone or methylprednisolone (corticosteroids)
  Interventions: Drug: Itacitinib (200 mg); Drug: prednisone or methylprednisolone (corticosteroids)
- Itacitinib (300 mg) (Experimental): Itacitinib (300 mg) + prednisone or methylprednisolone (corticosteroids)
  Interventions: Drug: Itacitinib (300 mg); Drug: prednisone or methylprednisolone (corticosteroids)

INTERVENTIONS:
Drug: Itacitinib (200 mg)
  Other Names: INCB039110
  Arms: Itacitinib (200 mg)
Drug: Itacitinib (300 mg)
  Other Names: INCB039110
  Arms: Itacitinib (300 mg)
Drug: prednisone or methylprednisolone (corticosteroids) — All subjects will receive prednisone 2.5 mg/kg per day PO (or methylprednisolone 2 mg/kg IV daily) on Days 1 through 5. Subjects will be tapered as tolerated beginning on Day 6 to no less than 0.25 mg/kg per day PO (or methylprednisolone 0.2 mg/kg per day) by Day 28. After Day 28, corticosteroids should be tapered according to institutional guidelines to attain ≤ prednisone 0.2 mg/kg per day (or ≤ methylprednisolone 0.16 mg/kg per day) by Day 56.

SUMMARY:
To determine if Itacitinib in combination with corticosteroids is safe and tolerable in patients with Grade IIB-IVD acute graft-versus-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Have undergone first allo-HSCT from any donor source (matched unrelated donor, sibling, haploidentical) using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative transplants are eligible.
* Clinically suspected Grades IIB to IVD acute GVHD as per modified MN-CIBMTR criteria, occurring after allo-HSCT with any conditioning regimen and any anti-GVHD prophylactic program.
* Subjects may, but are not required to, have previously received corticosteroids for acute GVHD:
* Evidence of myeloid engraftment. Use of growth factor supplementation is allowed.

Exclusion Criteria:

* Has received more than 1 hematopoietic stem cell transplantation.
* Has progressed on more than 2 prior treatment regimens for acute GVHD.
* Presence of an active uncontrolled infection.
* Subjects with relapsed primary disease, or subjects who have been treated for relapse after the allogeneic hematopoietic stem-cell transplantation (allo-HSCT) was performed.
* Inadequate recovery from toxicity and/or complications from the prior allo-HSCT.
* Any corticosteroid therapy (for indications other than GVHD) at doses > 1 mg/kg per day methylprednisolone or equivalent within 7 days of randomization.
* Previously received JAK inhibitor therapy for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of study treatment as measured by the frequency and severity of adverse events and serious adverse events | First dose of study drug to 30 days after the last dose of study drug

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Days 14, 28, 56 and 100
Maximum Observed Plasma Concentration (Cmax) of the two treatment groups Itacitinib | Day 1 and Day 7
Time to Reach the Maximum Plasma Concentration (Tmax) of the two treatment groups Itacitinib | Day 1 and Day 7
Area Under the Plasma Concentration-time Curve (AUC) of the two treatment groups Itacitinib | Day 1 and Day 7
Minimum observed plasma concentration (Cmin) of the two treatment groups Itacitinib | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (23):
- United States (23):
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Denver, Colorado
  - Coral Gables, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Westwood, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - San Antonio, Texas

REFERENCES:
- [Derived] Pratta M, Paczesny S, Socie G, Barkey N, Liu H, Owens S, Arbushites MC, Schroeder MA, Howell MD. A biomarker signature to predict complete response to itacitinib and corticosteroids in acute graft-versus-host disease. Br J Haematol. 2022 Aug;198(4):729-739. doi: 10.1111/bjh.18300. Epub 2022 Jun 11. PMID 35689489
- [Derived] Schroeder MA, Khoury HJ, Jagasia M, Ali H, Schiller GJ, Staser K, Choi J, Gehrs L, Arbushites MC, Yan Y, Langmuir P, Srinivas N, Pratta M, Perales MA, Chen YB, Meyers G, DiPersio JF. A phase 1 trial of itacitinib, a selective JAK1 inhibitor, in patients with acute graft-versus-host disease. Blood Adv. 2020 Apr 28;4(8):1656-1669. doi: 10.1182/bloodadvances.2019001043. PMID 32324888